CLINICAL TRIAL: NCT04373837
Title: An Innovative Rehabilitation Treatment of Time Deficits in Brain-damaged Patients Combining Prism Adaptation and Virtual Reality
Brief Title: Rehabilitation Treatment of Time Deficits in Brain-damaged Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ICS Maugeri CE 2194-Ob2A
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Brain Damage
Keywords: Right Brain Damaged Patients; Time perception; Mental Time Travel; Prismatic adaptation; Virtual Reality
MeSH Terms: conditions — Brain Injuries | interventions — Sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Without pre - With post (Experimental): Patients will perform two weeks treatment (10 sessions in total). First week: 5 days/week for 1 week, a daily session of pointing with neutral goggles inducing no-adaptation (NA) + Virtual Reality (VR) task (5 sessions).
  Second week: 5 days/week for 1 week, a daily session of pointing with prismatic goggles inducing prismatic adaptation (PA) + VR task (5 sessions).
  Interventions: Behavioral: Prismatic googles inducing prismatic adaptation (PA) associated to Virtual Reality (VR); Other: Neutral googles inducing no-adaptation (NA) associated to Virtual Reality (VR)
- Group 2: With pre - Without post (Experimental): Patients will perform two weeks treatment (10 sessions in total). First week: 5 days/week for 1 week, a daily session of pointing with prismatic goggles inducing prismatic (PA) + Virtual Reality (VR) task (5 sessions).
  Second week: 5 days/week for 1 week, a daily session of pointing with neutral goggles inducing no-adaptation (NA) + VR task (5 sessions).
  Interventions: Behavioral: Prismatic googles inducing prismatic adaptation (PA) associated to Virtual Reality (VR); Other: Neutral googles inducing no-adaptation (NA) associated to Virtual Reality (VR)

INTERVENTIONS:
Behavioral: Prismatic googles inducing prismatic adaptation (PA) associated to Virtual Reality (VR) — The experimental condition consists of PA procedure associated to VR task: the pointing task will be followed by 5 sessions of VR task.
  Pointing task. Patients will perform a session of 90 pointing movements toward a visual target presented in a variety of positions on the right, the left or at the center of the visual field. This pointing task will be performed with prismatic googles inducing a rightward shift of the visual field (experimental condition). After lenses removal, a leftward shift of spatial attention will be produced.
  Virtual Reality task consists of a 3D computer-generated virtual environment that will be displayed on a desktop VR computer monitor. A joystick will provide the graphical interface for patients by allowing user-friendly exploration of virtual scenarios. Patients will be presented 16 actions, with dynamic simulations of real life situations. They will verbally estimate and reproduce the duration of each previously presented action.
Other: Neutral googles inducing no-adaptation (NA) associated to Virtual Reality (VR) — The sham condition of this study consists of NA procedure associated to VR task: the pointing task will be followed by 5 sessions of VR task.
  Pointing task. Patients will perform a session of 90 pointing movements toward a visual target presented in a variety of positions on the right, the left or at the center of the visual field. This pointing task will be performed with neutral goggles (control condition), which should not induce a shift of the visual field and of spatial attention.
  Virtual Reality task consists of a 3D computer-generated virtual environment that will be displayed on a desktop VR computer monitor. A joystick will provide the graphical interface for patients by allowing user-friendly exploration of virtual scenarios. Patients will be presented 16 actions, with dynamic simulations of real life situations. They will verbally estimate and reproduce the duration of each previously presented action.

SUMMARY:
The efficacy of an innovative rehabilitation treatment for deficit in time processing is tested in right brain damaged patients.

Patients with a focal lesion following a stroke and without general cognitive impairment will be submitted to computerized tests assessing the ability to estimate time duration (intervals around 7500 ms) and to mental travel in time. Moreover, the impact of the deficit in time processing in everyday life will be evaluated by using ad hoc questionnaires.

Patients will perform tasks before and after two weeks of a new rehabilitation treatment, combining a training for one week with prismatic googles inducing prismatic adaptation (PA) plus Virtual Reality (VR) and a training for one week with neutral googles inducing no-adaptation (NA) plus Virtual Reality. Participants will be randomized into two groups. Each group will be submitted to both treatments in a different order, accordingly with a crossover design.

A greater amelioration in time processing after PA+VR than NA+VR training should be found. Moreover, an improvement in everyday life activities is expected accordingly with the amelioration in time processing.

DETAILED DESCRIPTION:
Time processing involves different abilities - i.e. estimating the duration of an event and moving in past and future time - and it is a fundamental ability in everyday life. However, in neuropsychology, time processing is routinely neglected in the assessment of cognitive deficits in brain-damaged patients. This is surprising since time is an important function that permeates our activities: we perceive mismatches in lip reading (milliseconds), we estimate how long it takes to be ready for work (minutes), and we plan how long it will take a manuscript to be accepted (usually months). Thus, impairment in processing time has important consequences in daily life.

For instance, it is known that right brain damaged (RBD) patients with spatial attentional deficit (neglect) are impaired in estimate the duration of a time interval as well as in the ability of mentally moving in time (Mental Time Travelling).

Previous studies have demonstrated an improvement of time estimation and mental time travel after a leftward shift of spatial attention induced by a single session of prismatic adaptation (PA). Moreover, a recent study investigated the long-term duration of the benefits induced by 10 daily sessions of PA treatment on mental time travel and functional abilities in neglect patients. Results suggest that the PA treatment induces a long-lasting and stable ameliorations of mental time travel and functional competences.

To generalize the effects of PA treatment to everyday life, here we propose to combine PA with a virtual reality training (VR). VR has recently been used as an effective tool both for the assessment and rehabilitation of cognitive deficits, because it allows post-stroke patients to interact with ecological environments similar to the real ones, but in a safe and controlled condition.

Aim of this study is to set up a rehabilitation procedure for temporal deficits, combining a well-established PA procedure with an innovative, more engaging and ecological VR approach.

Patients will perform tasks before and after two weeks of a new rehabilitation treatment, combining a training for one week with prismatic googles inducing prismatic adaptation (PA) plus Virtual Reality (VR) and a training for one week with neutral googles inducing no-adaptation (NA) plus Virtual Reality. Participants will be randomized into two groups. Each group will be submitted to both treatments in a different order, accordingly with a crossover design.

A greater amelioration in time processing after PA+VR than NA+VR training should be found. Moreover, an improvement in everyday life activities is expected accordingly with the amelioration in time processing.

ELIGIBILITY:
Inclusion Criteria:

* patients with focal right brain-damage

Exclusion Criteria:

* generalized cognitive impairment (score lower than 24 at the Mini Mental State Examination)
* psychiatric disorders
* additional neurological disorders
* abusive use of alcohol or illicit drugs

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Change in Mental Time Travel Ability on the Mental Time Travel (MTT) Task | baseline, after one week treatment (T1), after two weeks treatment (T2), one week after the end of treatment (follow-up)
  In the MTT task participants are listened to auditory stimuli consisting of brief descriptions of personal and non-personal events. They are required to project themselves in the past (10 years ago), present or future (10 years from now) and to verbally determine whether each event has already happened (relative past event) or is yet to happen (relative future event) with respect to the specific self-location in time (past, present and future).
  Error rates and reaction times will be recorded and analyzed. The improvement will be defined as changes in the Inverse Efficiency (IE) ability: reaction times/accuracy.
Change in Time Estimation Ability on the Time Estimation Task | baseline, after one week treatment (T1), after two weeks treatment (T2), one week after the end of treatment (follow-up)
  The Time Estimation task consists of a red square that is displayed for different durations (3500, 5500, 7500, 9500, 11500 ms) on the computer screen. Participants are instructed to verbally judge whether the duration of each stimulus is "short" or "long" with respect to previously acquired pair of reference durations (3500 and 11500 ms).
  A psychophysical response function will be created for each participant by calculating the proportion of "long" responses: the Point of Subjective Equality (PSE) is the duration at which a participant is equally likely to classify the stimuli as short or long. An increase of "long" response after treatment, as compared to baseline performance, induces a decreased PSE, reflecting a relative shift towards overestimation of temporal midpoint. Conversely, an increase of "short" responses after treatment, as compared to baseline performance, induces an increased PSE, reflecting a relative shift towards underestimation of temporal midpoint.
Change in Time Reproduction Ability on the Time Reproduction Task | baseline, after one week treatment (T1), after two weeks treatment (T2), one week after the end of treatment (follow-up)
  In the Time Reproduction task a blue square is presented for a variable time interval (3500, 5500, 7500, 9500, 11500 ms) on the computer screen. Next, a red square appears on the screen and participants are instructed to reproduce the entire duration of the preceding blue square by pressing the space bar on the keyboard.
  For each subject, the reproduced time intervals before PA will be subtracted from the reproduced time intervals after PA. Thus, this difference will be positive when reproduced time will be longer after than before treatment (underestimation of time duration) and negative when reproduced time will be shorter after than before treatment (overestimation of time duration).

SECONDARY OUTCOMES:
Assessment of General Cognitive Functioning on the Mini Mental State Examination (MMSE) | baseline
  The MMSE is a 30-point questionnaire that examines functions including registration (repeating named prompts), attention and calculation, recall, language, ability to follow simple commands and orientation. The score ranges from 0 to 30 (cut-off = 24).
Assessment of Verbal Comprehension on the Token Test | baseline
  The Token Test is a test of auditory language processing in which participants are asked to manipulate tokens of different shapes, sizes, and colors in response to increasingly complex instructions. One point is credited for a correct performance on the first presentation and 0.5 point if the performance is correct only on the second presentation. The score ranges from 0 to 36 (cut-off = 26,50).
Assessment of Unilateral Spatial Neglect on the Behavioral Inattention Test (BIT) | baseline
  The BIT is composed of two scales, the Conventional scale and the Behavioral scale. Participants will be administered the Conventional scale, which includes 6 tasks: line crossing, letter cancellation, star cancellation, figure and shape copying, line bisection and representational drawing. The score ranges from 0 to 146 (cut-off = 129).
Assessment of Frontal Functions on the Wisconsin Card Sorting Test (WCST) | baseline
  In the WCST, people have to classify cards according to different criteria. There are four different ways to classify each card, and the only feedback is whether the classification is correct or not. The classification rule changes every 10 cards. Three scores will be calculated: global score, perseveration errors and non-perseveration errors. The global score is computed by subtracting from the total number of administered trials the number of categories completed multiplied by ten = [n° of trials - (n° of achieved categories x 10)].
  The score ranges from 128 to 0, i.e. the lower the score, the better the performance.
Assessment of Memory on the Rey's 15 Words Auditory Learning Test | baseline
  The test is designed as a list-learning paradigm in which the participant hears a list of 15 nouns and is asked to recall as many words from the list as possible (five repetitions of free-recall). After a 15 min delay, the participant is asked to again recall the words from the list. It provides two scores: immediate (range 0-75) and delayed recall (range 0-15), i.e. the higher the score, the better the performance.
Change in Unilateral Spatial Neglect on the Bells Cancellation Test | baseline, after two weeks treatment (T2), one week after the end of treatment (follow-up)
  The subject is required to cross out the bells that are scattered among several different shapes on a sheet of paper. Two indices of neglect will be calculated: total number of omissions (cut-off < 5) and number of left omissions (cut-off < 5), i.e. the difference between the number of targets crossed out on the right side and the number of targets crossed out on the left side (asymmetry score).
Change in Unilateral Spatial Neglect on the Apples Cancellation Test | baseline, after two weeks treatment (T2), one week after the end of treatment (follow-up)
  This is a cancellation task in which outline drawings of 150 apples are shown pseudorandomly scattered over a sheet of A4 paper presented in a landscape orientation. All of the apples are presented in an upright position. One-third of the apples are full (targets) and two-thirds are open on either the left or the right side (distractors). Participants are asked to cross out all the full apples and to ignore the distractors. Three scores will be calculated: full apples barrage (cut-off = 45), full apples asymmetry (cut-off = 2), and incomplete apples asymmetry (cut-off = 1).
  The full apples asymmetry (the difference between the number of targets selected on the right side and the number of targets selected on the left side) represents the score for egocentric neglect. The incomplete apples asymmetry (total left openings minus total right openings) represents the score for allocentric neglect.
Change in Frontal Functions on the Frontal Assessment Battery (FAB) | baseline, after two weeks treatment (T2)
  The FAB is a brief battery of six neuropsychological tasks designed to assess frontal lobe function at bedside. The six tasks explore: conceptualization and abstract reasoning, lexical verbal fluency and mental flexibility, motor programming and executive control of action, self-regulation and resistance to interference, inhibitory control, and environmental autonomy.
  Each task scores from 0 (pathologic) to 3 (best performance), for a total maximum score of 18.
Change in Verbal Estimation Ability on the Time and Weight Estimation Test (STEP) | baseline, after two weeks treatment (T2)
  The STEP assesses aspects of executive functioning related to cognitive estimation ability. The questionnaire is composed of two distinct ten-item sections, focusing on time (e.g., How long does it take to have a shower?) and weight (e.g., How heavy is a pair of jeans?) estimations. Each item scores from 0 (bizarre estimation) to 3 (best estimation), for a total maximum score for each section of 30, with a cut-off value for normality above 20 for each section.
Change in Verbal Estimation Ability on the Cognitive Estimation Task (CET) | baseline, after two weeks treatment (T2)
  The test comprised 21 questions that required participants to give oral, numerical responses. Two different scoring procedures will be considered: absolute error score and bizarreness. The total score for all 21 items ranges from a best of zero to a worst of 42. The greater the error score, the poorer the performance on the CET (cut-off = 18). The total bizarreness score ranges from 0 and 21 (cu-off = 4). The higher the bizarreness score, the greater the impairment in cognitive estimation.
Change in Functional Abilities on the Questionnaire of Temporal Ability | baseline, after two weeks treatment (T2), one week after the end of treatment (follow-up)
  The Questionnaire of temporal ability is a new instrument to measure the ability to locate daily activities in time.
Change in Functional Abilities on the Motricity Index | baseline, after two weeks treatment (T2)
  The Motricity Index is a standardized mobility scale, designed to measure the motor impairment of the trunk and the right and left upper and low limbs. Each component part of the index expresses the strength of the part of the body that is evaluated. The score ranges from 0 (low motor functions) to 100 (high motor functions).
Change in Functional Abilities on the Activities of Daily Living (ADL) | baseline, after two weeks treatment (T2), one week after the end of treatment (follow-up)
  Eleven ADL areas, such as walking, dressing, cleaning, and feeding, are assessed to measure the degree of independence in activities of daily living. Each activity is evaluated through a 5-points questionnaire (1 = completely independent, 5 = completely dependent), with a total score ranging from 11 (high independence in ADL) to 55 (high dependence in ADL).
Change in Functional Abilities on the Functional Independent Measure (FIM) | baseline, after two weeks treatment (T2)
  The FIM is an 18-item, 7-level scale developed to uniformly assess severity of patient disability and medical rehabilitation functional outcome. Scores range from 18 (lowest) to 126 (highest) indicating level of function.
Change in Spatial Working Memory on the Spatial Working Memory Test | baseline, after two weeks treatment (T2)
  Participants are presented with a paper sheet composed of 24 identical Os and 24 different drawings of common objects and they are instructed to cancel all Os, marking each once only. The score is the number of re-cancellations, that will be scored for any additional cross (an extra single line is scored as 0.5 re-cancellation).

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Frassinetti, PhD, Principal Investigator — Istituti Clinici Scientifici Maugeri IRCCS
Locations (1):
- ICS Maugeri IRCCS, U.O. di Rieducazione e Recupero funzionale di Castel Goffredo, Castel Goffredo, Mantova, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anelli F, Avanzi S, Arzy S, Mancuso M, Frassinetti F. Effects of spatial attention on mental time travel in patients with neglect. Cortex. 2018 Apr;101:192-205. doi: 10.1016/j.cortex.2018.01.012. Epub 2018 Feb 2. PMID 29482017
- [Background] Anelli F, Avanzi S, Damora A, Mancuso M, Frassinetti F. Mental time travel and functional daily life activities in neglect patients: Recovery effects of rehabilitation by prism adaptation. Cortex. 2019 Apr;113:141-155. doi: 10.1016/j.cortex.2018.12.003. Epub 2018 Dec 14. PMID 30660953
- [Background] Appollonio I, Leone M, Isella V, Piamarta F, Consoli T, Villa ML, Forapani E, Russo A, Nichelli P. The Frontal Assessment Battery (FAB): normative values in an Italian population sample. Neurol Sci. 2005 Jun;26(2):108-16. doi: 10.1007/s10072-005-0443-4. PMID 15995827
- [Background] Carlesimo GA, Caltagirone C, Gainotti G. The Mental Deterioration Battery: normative data, diagnostic reliability and qualitative analyses of cognitive impairment. The Group for the Standardization of the Mental Deterioration Battery. Eur Neurol. 1996;36(6):378-84. doi: 10.1159/000117297. PMID 8954307
- [Background] De Renzi E, Faglioni P. Normative data and screening power of a shortened version of the Token Test. Cortex. 1978 Mar;14(1):41-9. doi: 10.1016/s0010-9452(78)80006-9. PMID 16295108
- [Background] Della Sala S, MacPherson SE, Phillips LH, Sacco L, Spinnler H. How many camels are there in Italy? Cognitive estimates standardised on the Italian population. Neurol Sci. 2003 Apr;24(1):10-5. doi: 10.1007/s100720300015. PMID 12754651
- [Background] Demeurisse G, Demol O, Robaye E. Motor evaluation in vascular hemiplegia. Eur Neurol. 1980;19(6):382-9. doi: 10.1159/000115178. PMID 7439211
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Frassinetti F, Magnani B, Oliveri M. Prismatic lenses shift time perception. Psychol Sci. 2009 Aug;20(8):949-54. doi: 10.1111/j.1467-9280.2009.02390.x. Epub 2009 Jun 22. PMID 19549081
- [Background] GRANT DA, BERG EA. A behavioral analysis of degree of reinforcement and ease of shifting to new responses in a Weigl-type card-sorting problem. J Exp Psychol. 1948 Aug;38(4):404-11. doi: 10.1037/h0059831. No abstract available. PMID 18874598
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Laiacona M, Inzaghi MG, De Tanti A, Capitani E. Wisconsin card sorting test: a new global score, with Italian norms, and its relationship with the Weigl sorting test. Neurol Sci. 2000 Oct;21(5):279-91. doi: 10.1007/s100720070065. PMID 11286040
- [Background] Linacre JM, Heinemann AW, Wright BD, Granger CV, Hamilton BB. The structure and stability of the Functional Independence Measure. Arch Phys Med Rehabil. 1994 Feb;75(2):127-32. PMID 8311667
- [Background] Mancuso M, Rosadoni S, Capitani D, Bickerton WL, Humphreys GW, De Tanti A, Zampolini M, Galardi G, Caputo M, De Pellegrin S, Angelini A, Bartalini B, Bartolo M, Carboncini MC, Gemignani P, Spaccavento S, Cantagallo A, Zoccolotti P, Antonucci G. Italian standardization of the Apples Cancellation Test. Neurol Sci. 2015 Jul;36(7):1233-40. doi: 10.1007/s10072-015-2088-2. Epub 2015 Jan 25. PMID 25618236
- [Background] Oliveri M, Magnani B, Filipelli A, Avanzi S, Frassinetti F. Prismatic adaptation effects on spatial representation of time in neglect patients. Cortex. 2013 Jan;49(1):120-30. doi: 10.1016/j.cortex.2011.11.010. Epub 2011 Nov 27. PMID 22200531
- [Background] Patane I, Farne A, Frassinetti F. Prismatic Adaptation Induces Plastic Changes onto Spatial and Temporal Domains in Near and Far Space. Neural Plast. 2016;2016:3495075. doi: 10.1155/2016/3495075. Epub 2016 Feb 14. PMID 26981286
- [Background] Pedroli E, Serino S, Cipresso P, Pallavicini F, Riva G. Assessment and rehabilitation of neglect using virtual reality: a systematic review. Front Behav Neurosci. 2015 Aug 25;9:226. doi: 10.3389/fnbeh.2015.00226. eCollection 2015. PMID 26379519
- [Background] Wilson B, Cockburn J, Halligan P. Development of a behavioral test of visuospatial neglect. Arch Phys Med Rehabil. 1987 Feb;68(2):98-102. PMID 3813864
- [Background] Wojciulik E, Husain M, Clarke K, Driver J. Spatial working memory deficit in unilateral neglect. Neuropsychologia. 2001;39(4):390-6. doi: 10.1016/s0028-3932(00)00131-7. PMID 11164877